CLINICAL TRIAL: NCT04297761
Title: Cardiovascular Effects of Exposure to Wood Smoke in Healthy Human Adults
Acronym: MASKOFF
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: MASKOFF has been suspended while the study activities are transferred from the EPA Human Studies Facility in Chapel Hill to the EPA Office of Research and Development headquarters at Research Triangle Park.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-2078
Record Dates: First submitted 2020-02-27; First posted 2020-03-05 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Healthy
Keywords: Healthy subjects; Wood smoke; Respiratory effects; Cardiovascular effects; Young

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Controlled Exposure (Experimental): All subjects will be exposed to both air containing wood smoke and filtered air for 2 hours with alternating 15 minutes of exercise (cycle ergometer) and rest.
  Interventions: Other: Filtered Air; Other: Wood Smoke

INTERVENTIONS:
Other: Filtered Air — Ambient air will be filtered and used for control exposure.
Other: Wood Smoke — Wood smoke is generated by smoldering dry white oak logs and the exposure level will be maintained at an average of 500 µg/m^3 for 2 hours.

SUMMARY:
MASKOFF Clinical Trials 8/22/23

Brief Summary:

Purpose: The study is designed to investigate cardiovascular effects of young healthy human subjects exposed to wood smoke.

Participants: Approximately 80 young (18-35 years old) healthy subjects to complete.

Procedure (methods): After consenting to participate in the study, subjects will be exposed first to filtered air and on the next exposure day to approximately 500 µg/m^3 wood smoke. Both exposures will be 2 hours long with alternating 15 min of exercise (cycle ergometer) and 15 min rest period. The exercise level will be adjusted to achieve approximately 20 L/min/m^2 minute ventilation. Venous blood samples and measurements of lung, cardiac and vascular function will be made prior to and immediately following each exposure. Induced sputum samples and nasal epithelial lining fluid will be collected approximately 24 hours post each exposure.

DETAILED DESCRIPTION:
Wood smoke pollution is a common problem across the world, including in the US. This wood smoke comes from people using wood to heat and cook, as well as from wildfires. The purpose of this research study is to investigate the cardiovascular effects of exposure to wood smoke in young, healthy human subjects. Results from this study will also increase understanding of how wood smoke exposure adversely affects the functioning of the human cardiovascular and respiratory systems. This understanding may be especially important for patients with cardiopulmonary diseases.

There is a likelihood that due to scheduling conflicts and other unexpected scenarios (such as government shutdowns etc.) that the time between consenting and participation could be delayed, although every effort will be made to accommodate subjects without hurting the integrity of the study. There will be 5 sessions, including a consenting session which will last for about 5 hours. The two exposure-day sessions will last approximately 8-9 hours each and will occur 48 hours apart. There will also be two follow-up visits lasting approximately 4-hours each on the day following the participants' last exposure.

Before consenting to be part of this study, the potential participant must read all consent forms in entirety. The research and medical staff will then answer all of the participants' questions and explain the risks involved in this study to satisfaction.

The participant should have already undergone a general physical examination to ensure that said participant is a suitable candidate for this study. Participants who were assigned female at birth will be asked about menstrual history and a pregnancy test will be performed. This will be repeated on each exposure day if more than 7 days have lapsed since the last pregnancy test at the HSF.

Consenting Day:

The consent day visit is expected to last about 4-5 hours. The investigators will review the inclusion and exclusion criteria and the participants' medical conditions and current medications. The investigators will go over the study in detail so the participant is as informed as possible before consenting to being part of this study. The participant will then sign all consent forms and receive one set of signed copies. The participant will also tour the exposure chambers following the consenting process. After consenting, the participant's vital signs and approximately 4 ml of blood will be collected. This blood will be measured for specific analytes to ensure the participant can safely complete the study.

The participant will perform a breathing test (spirometry) to measure lung function. The participant will breathe through a filter into a plastic tube, while being coached by members of the study team. Participants will be asked to take a full breath in, follow by a hard and fast maximal exhalation. The participant will be asked to do this several times. This test measures the volume of air that can be exhaled and the rate of airflow during exhalation after a maximal inhalation. This is a method to measure lung function which must meet certain criteria (lung capacity and volume) prior to exposure in order for the participant to remain in the study. Lung function test results should be equal to or greater than 80% of the reference value to continue participation in the study.

As part of the consenting day, participants will undergo exercise training to determine the level of exercise needed to reach the target minute ventilation for this study. Participants will pedal on an exercise bike at various levels of resistance for 5-15 minute periods while minute ventilation (how much air is being inhaled per minute) is measured at regular intervals using a mouthpiece tachometer. Displacement bands will be placed around the participants' torso to measure minute ventilation via chest expansion while exercising.

Participants will also undergo procedures for nasal epithelial lining fluid sampling (nasal mucosa) and induced sputum collection. It is known that less than half of normal, healthy people can produce a sputum sample that is of acceptable quality for analysis. The study will end if a participant is a non-producer or the quality of the sputum produced does not meet the study inclusion criteria. In this event, the participant will be reimbursed for the consenting session.

Participants who meet all inclusion criteria will be contacted with further instructions.

It may be possible to reschedule in the event of severe weather, the participant becomes ill (for example, a cold or respiratory infection), or other unforeseen circumstances.

Exposure days:

The study team will contact and send reminders to all participants a few days before the exposure session. Participants should avoid smoke, fumes, alcohol, and strenuous exercise 24 hours prior to all visits, and abstain from pan fried or grilled meat after midnight of the exposure day.

Participants will be asked to eat a light breakfast and arrive at the EPA medical station by 8:00 am. The study team will make ensure that all participants understand the importance of arriving earlier to ensure the investigators have adequate time to process all samples and data. Participants who arrive after 8:00 am will be unenrolled from the study.

Prior to exposure, a study team member will collect the follow from each participant:

1. Vital signs (heart rate, respiratory rate, blood pressure, oxygen saturation level) and an electronic symptom questionnaire.
2. Heart Rate Variability via a Holter monitor. A study team member will attach ten electrocardiogram (ECG) leads to the participants' chest. It may be necessary to clean and shave areas of the chest where these leads will be placed. Participants will be asked to not apply excessive deodorant, skin lotions, and body sprays on as these may interfere with data recording. The leads will be connected to 2 monitors (small recording devices about the size and weight of a cell phone) to obtain heart rate and rhythm readings. It is preferable that the electrodes will stay in place for approximately 4 days as these measurements will be collected several times during the study, however, participants will be given the option to remove the electrodes by the end of each exposure day. To begin recording, participants will be asked to recline quietly for 30 minutes. It is important that the participant does not fall asleep during this 30-minute period. These measurements will allow the investigators to determine whether wood smoke exposure causes small changes in the ability of your nervous system to regulate how your heart beats.
3. Retinal Imaging. An ophthalmic camera will be employed to collect retinal images of all participants before and after each exposure and on the follow-up visit. The participants chin will be rested in front of the camera, while a study team member takes pictures of both eyes. Glasses or contacts must be removed for this test. Participants will be notified to bring contact lens cases and solutions.
4. The study team will continue to store the images for future undesignated studies given the participant's consent. This allows the team to make the best use of the images collected from subjects. Participants will be given a separate consent form for this storage and do not have to allow images to be stored indefinitely in order to participate in this study.
5. Blood Draw. Approximately 30 mL of blood will be drawn (about 2 tablespoons) on the train day, before and after each exposure and on the follow-up visit. The study team will test this blood to see blood cell function is affected by exposure to wood smoke. A small portion of the blood sample will be used to measure the relative content of various fatty acids present in blood. With permission, the investigators will also store some of the blood obtained during the study for yet-to-be-determined tests.
6. Spirometry will be performed following the same procedure used on the consent day.
7. Ventilation Rate. BioPac bands will be placed around the participants' thorax and abdomen. These bands will be connected to a monitor that wirelessly transmits readings of breathing volume and rate. These measurements will allow the investigators to determine if the participants' exercise workload is sufficient to meet the study's target minute ventilation rate.

Participants will enter the exposure chamber following the pre-exposure protocol listed above. While in the chamber, participants will undergo exposure for 2 hours of either clean filtered air or wood smoke. Participants will receive clean filtered air on one day and wood smoke on the other day. Subjects will be blinded as to which exposure they receive on each exposure day. The concentration of wood smoke that used in this study (approximately 500 μg/m^3) is below what someone would be exposed to during biomass burning for heating and food preparation or in the surrounding area of a forest fire or agricultural burning. Chamber conditions will be at a comfortable temperature and relative humidity. Participants will perform mild exercise on a stationary bicycle in the chamber every other 15 minutes alternating with resting period for a total of 1 hour of exercise per chamber exposure. The target ventilation rate will be maintained at approximately 20 L/min/m^2 and monitored using a pneumotach and the BioPac bands. A study coordinator or other trained person will be observing from outside the chamber at all times. During the exposure, heart rate and oxygen saturation will be monitored by placing a device (pulse oximeter) on the participants' finger. If it appears the participant is experiencing significant discomfort, breathing or heart problems, the exposure will be terminated immediately. In addition, the participant may elect to terminate the exposure at any time for any reason. Participants who do not complete the study protocol will be fully compensated that day's session but will be ineligible for further participation in the study.

Immediately following the exposure, participants will:

1. Fill out a symptom score questionnaire electronically.
2. Have your vital signs checked.
3. Have blood drawn (Approximately 30 mL, about 2 tablespoons).
4. Have a breathing test (spirometry).
5. Recline quietly for 30 minutes while heart rhythm is recorded.
6. Have retinal pictures will be taken.
7. Eat a low-fat lunch brought from home. At this time, the study team will encourage participants to take a shower in a private shower facility at the HSF to get rid of the wood smoke odor. Towel, soap, and shampoo will be provided. The participant's belongings will be securely stored during all visits.

Participants will be assessed and discharged by the study team following the completion of each exposure day.

Follow up visit (about 4 hours):

Participants will return to the HSF the next morning (approximately 24 hours after exposure) and will:

1. Have vital signs checked.
2. Recline quietly for 30 minutes while your heart rhythm is recorded. Electrodes will be removed from the participants' chest at the end of this test.
3. Have blood pressure and heart rate measured.
4. Fill out a symptom score questionnaire electronically.
5. Complete TracMyAir Questionnaire (see below)
6. Have NELF samples collected.
7. Have samples of induced sputum collected.
8. Have a breathing test (spirometry).
9. Have blood drawn (approximately 30 mL) for analysis.
10. Have retinal pictures taken.

TracMyAir is an application that uses data from nearby monitoring stations to report on local air pollution levels. The study team will use TracMyAir to determine each study participant's daily (24 hour average) ambient PM2.5 and ozone exposure and inhaled dose. TracMyAir calculates daily 24 hour average exposure and dose for the previous 4 days, which allows for a lag analysis. TracMyAir uses EPA's previously developed and evaluated Exposure Model for Individuals (EMI). The EPA staff will enter input data (shown below) into the TracMyAir software for each study participant.

If there are any samples left over after all study information is collected, the study team will continue to store the samples for future undesignated studies given the participant's consent. This allows the team to make the best use of the samples collected from subjects. Participants will be given a separate consent form for this storage and do not have to allow samples to be stored indefinitely in order to participate in this study.

ELIGIBILITY:
Inclusion criteria:

1. Age 18-35 years old , healthy, with a Body Mass Index (BMI, kg/m^2) values ≥ 19 and ≤ 34, inclusive).
2. Physical conditioning that allows intermittent, mild exercise for approximately 60 min during a 2 hour exposure session. The volunteer must be able to complete the exposure exercise regimen at a workload sufficient to induce a minute ventilation rate of approximately 20 L/min/m^2 for 15 min without exceeding 80% of projected maximal heart rate.
3. Normal ECG.
4. Normal lung function based on NHANES III reference values. i. Forced vital capacity (FVC) ≥ 80% of that predicted for age, gender, ethnicity, and height.

   ii. Forced expiratory volume in one second (FEV1) ≥ 80% of that predicted for age, gender, ethnicity, and height.

   iii: FEV1/FVC ratio ≥ 70% (absolute value)
5. Oxygen saturation greater than 94% at the time of physical exam.

Exclusion criteria:

1. Individuals with the following conditions:

   * A history of acute or chronic cardiovascular disease, chronic respiratory disease, cancer, rheumatologic disease, neuromuscular disease, or immunodeficiency state.
   * BMI (kg/m^2) values < 19 and > 34.
   * Blood pressure readings ≥ 140 systolic and/or ≥ 90 diastolic.
   * Diabetes (previously diagnosed or with hemoglobin A1c level equal to or greater than 6.4%).
   * Asthma or a history of asthma.
   * Bleeding/clotting disorders.
2. Individuals with a cardiovascular disease risk score greater than 10% using the ACC/AHA ASCVD risk calculator. (Based on the 10-year risk of heart disease or stroke using the Atherosclerotic Cardiovascular Disease algorithm published in 2013 American College of Cardiology/American Heart Association Guideline on the Assessment of Cardiovascular risk.)
3. Individuals who have unspecified illnesses, which in the judgment of the medical staff might increase the risk associated with wood smoke inhalation will be a basis for exclusion.
4. Individuals who have had recent (within 6 months) abdominal an/or eye surgery, or with any types of hernia, as well as any other contraindicators for raised intra-abdominal pressure.
5. Individuals who are currently taking systemic steroids or oral anticoagulants long term.
6. Individuals who are taking prescribed medications such as ß-blocker medications, that may impact the results of wood smoke challenge for the duration of the study. Other medications not specifically mentioned here may be reviewed by the medical staff prior to an individual's inclusion in the study. Use of other medications will be evaluated on a case-by-case basis. There is the potential that an individual's current medication use will preclude them from participating in the study at the current time, but they may be reassessed and potentially rescheduled for participation later based on the judgement of the medical staff.
7. Individuals who are allergic to:

   * Chemical vapors or gases.
   * Tape or electrodes on their skin.
   * Or individuals with active allergies or currently experience allergy related symptoms
8. Individuals who are pregnant, attempting to become pregnant or breastfeeding.
9. Individuals who are currently smoking (including vaping, hookah and e-cigarette) or have smoking history within 1 year of study or have an equal to greater than or a 5-pack year smoking history.
10. Individuals living with a smoker who smokes inside the house.
11. Individuals who are regularly exposed to high levels of vapors, dust, gases, or fumes.
12. Individuals who do not read, speak, or understand English well enough to give informed consent.
13. Individuals that are unable to perform the exercise required for the study.
14. Individuals who are unwilling or unable to stop taking any current dietary supplements or vitamins for the duration of the study.
15. Individuals currently taking prebiotics, probiotics, or antihistamines.
16. Individuals who have experienced an acute respiratory illness within the last 6 weeks.
17. Individuals that will NOT comply with the following requirements:

    * Avoid smoke and fumes for 24 hours before all visits.
    * Avoid exposure to unvented household combustion sources (gas stoves, lit fireplaces, oil/kerosene heaters) for 48 hours before all visits.
    * Avoid over-the-counter pain medications such as aspirin, Advil, Aleve, or NSAIDs for 48 hours before all visits.
    * Avoid drinking alcohol 34 hours before all visits
    * Avoid strenuous exercise for 24 hours prior to an after all visits.
    * Eat a light breakfast and low-fat lunch on the exposure day.
    * Refrain from eating pan fried and/or grilled foods 12 hours prior to the exposure days.
    * Refrain from consuming caffeine for 12 hours prior to all study visits.
    * Refrain from consuming food 2 hours prior to the consenting and follow up sessions, as this may interfere with induced sputum collection.
    * Wear a N95 mask during all visits to the HSF. A mask will be provided to participants upon check-in.

Since examining changes of cells in the induced sputum is an important test for this study, if a subject is a non-producer, or if the quality of their sputum sample does not meet the requirements, they will be disqualified and imbursed for participation up to this point.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in polymorphonuclear neutrophils (PMN%) in the Sputum | Day 1, Day 3, Day 5
  Airway inflammation will be assessed by the % PMN in the sputum

SECONDARY OUTCOMES:
Change in Forced Expired Volume in the First Second (FEV1) (liter) | Day 1, Day 2, Day 3, Day 4, Day 5
  FEV1 is determined by spirometry
Change in Forced Vital Capacity (FVC) (liter) | Day 1, Day 2, Day 3, Day 4, Day 5
  FVC is determined by spirometry
Change in Diameters (mm) of Retinal Arteries and Veins | Day 2, Day 3, Day 4, Day 5
  Retinal images will be taken using an FDA-approved, commercially available, non-mydriatic fundus camera. Images will be taken from both eyes.
Percent Change in Heart Rate Variability | Day 2, Day 3, Day 4, Day 5
  Heart rate variability will be collected by the Holter monitor recording.
Change in Blood Fatty Acids (ng/mL) | Day 2, Day 3, Day 4, Day 5
  Blood sample will be collected for fatty acids analysis.
Change in Blood Cholesterol (ng/mL) | Day 2, Day 3, Day 4, Day 5
  Blood sample will be collected for blood cholesterol analysis.
Change in Cytokines in Nasal Epithelial Lining Fluid (NELF) (ng/mL) | Day 1, Day 2, Day 3, Day 4, Day 5
  NELF samples will be collected for cytokine measurements.
Change in interleukin-6, interleukin-8, interleukin-1 beta, and tumor-necrosis factor alpha in blood. (pg/mL) | Day 2, Day 3, Day 4, Day 5
  Blood will be collected prior to and post exposure to analyze for inflammatory markers.
Change in C-reactive protein in blood. (mg/dL) | Day 2, Day 3, Day 4, Day 5
  Blood will be collected prior to and post exposure to analyze for inflammatory markers.

CONTACTS AND LOCATIONS:
Overall Officials: James Samet, PhD, Principal Investigator — Environmental Protection Agency (EPA)
Locations (1):
- U.S. Environmental Protection Agency Human Studies Facility, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data will be shared through the U.S. EPA's ScienceHub database. ScienceHub is used to upload and store datasets associated with journal articles. Non-sensitive datasets are then made publicly accessible via the Environmental Dataset Gateway in fulfillment of the EPA's requirement to adhere to the Office of Management and Budget's Open Data Policy.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be available to the public after the conclusion of the study and the publication of the manuscripts.
Access Criteria: Data will be available at the U.S. EPA Science Hub.
URL: https://catalog.data.gov/dataset/epa-sciencehub